CLINICAL TRIAL: NCT03781973
Title: Bridging the Gap to Optimize Care and Outcomes for Youth With Diabetes Between Pediatric and Adult Diabetes Care
Brief Title: Bridging the Gap to Adult Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rayzel Shulman, Scientist Track Investigator, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CTO project ID: 1581
Record Dates: First submitted 2018-12-13; First posted 2018-12-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Type1diabetes
Keywords: Transition to adult care; Glycemic control

STUDY DESIGN:
Intervention Model Description: An intervention with integrated components
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pre-intervention (No Intervention): Those whose last pediatric visit was in the year before the intervention (2018).
  Medical record data abstracted from patient charts at the time of the final pediatric visit.
- Early Intervention (Other): Those whose last pediatric visit was in the year immediately after the start of the intervention (2019).
  The intervention will begin on Jan 1, 2019 and includes the following :
  1. Data Platform: Medical record data abstracted from patient charts at the time of the final pediatric visit. .
  2. Quality performance feedback reports: We will generate centre-level performance reports. Centres will be able to compare their performance to that of all other centres and to achievable benchmarks.
  3. Patient transition experience surveys at the final pediatric visit and 12 months later.
  4. Diabetes teams may direct patients and families to online transition resources.
  Interventions: Behavioral: Data platform +Quality Performance feedback reports
- Post-Intervention (Other): Those whose last pediatric visit was in the second year after the intervention (2020).
  The intervention includes the following :
  1. Data Platform: Medical record data abstracted from patient charts at the time of the final pediatric visit. .
  2. Quality performance feedback reports: We will generate centre-level performance reports. Centres will be able to compare their performance to that of all other centres and to achievable benchmarks.
  3. Patient transition experience surveys at the final pediatric visit and 12 months later.
  4. Diabetes teams may direct patients and families to online transition resources.
  Interventions: Behavioral: Data platform +Quality Performance feedback reports

INTERVENTIONS:
Behavioral: Data platform +Quality Performance feedback reports — Teams from each of the participating sites will attend the webinars. Each site will share an example of a QI initiative that they are executing and describe the success and challenges.
  Arms: Early Intervention; Post-Intervention

SUMMARY:
Adolescents with type 1 diabetes face particular challenges related to having a chronic illness that requires daily intensive self-management and medical follow-up during a period when their social, developmental, educational, and family situations are in flux. When transitioning from pediatric to adult care, over a third of youth have a care gap of >6 months. During this vulnerable period youth are at risk for acute life-threatening complications such as diabetic ketoacidosis, and for poor glycemic control, which confers an increased risk of chronic diabetes complications. Gaps in care may be a result of deficiencies in transition processes causing some young people to be poorly prepared for adult care and dissatisfied with the transition process. Ineffective transition can lead to decreased frequency of diabetes visits and an increased risk of adverse events in young adulthood. Further, risk factors such as psychiatric comorbidity and behavioural problems in adolescents with type 1 diabetes are associated with poor outcomes in early adulthood. Quality improvement initiatives can be designed to optimize care processes such as referral systems to adult diabetes providers.

Our overall objective is to optimize care and outcomes for youth with diabetes as they transition to adult care.

Specific Aim 1: To improve glycemic control in youth around the time of transition from pediatric to adult diabetes care Specific Aim 2: To evaluate the fidelity and quality of a quality improvement intervention designed to improve transition care processes and to identify contextual factors associated with variation in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All youth with a clinical diagnosis of type 1 diabetes followed at participating centres at the time of their final pediatric clinic visit between Jan 1, 2018 and Dec 31, 2020.
* Participants will be transitioning to Adult Care (ages ~16-19 yrs).
* Capacity to read and understand English (we estimate that >95% of participants will fulfill this requirement).
* Capacity to consent for themselves.

Exclusion Criteria:

* Individuals with non-type 1 diabetes.
* Individuals with type 1 diabetes who move out of Ontario within 12 months after their final pediatric visit.
* Individuals with type 1 diabetes who do not have the capacity to consent for themselves.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 484 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c | HbA1c value up to 12 months after the final pediatric visit.
  Hemoglobin A1c

SECONDARY OUTCOMES:
Number of Diabetes-related admissions, ED visits, death | number of occurrences up to12 months after the final pediatric visit.
  The occurrence of at least one diabetes-related admissions or emergency department visit or death
Time from the final pediatric visit to the first adult diabetes visit | Time in months up to 12 months after the final pediatric visit
  identified using physician service claims and defined as the first diabetes office visit by an adult endocrinologist, internist, or family physician

CONTACTS AND LOCATIONS:
Overall Officials: Rayzel Shulman, Md, PhD, Principal Investigator — The Hospital for Sick Children
Locations (5):
- Canada (5):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital, London Health Sciences Centre, London, Ontario
  - Markham Stouffville Hospital, Clinic 4, Markham, Ontario
  - Trillium Health Partners, Mississauga, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmad SZ, Ivers N, Zenlea I, Parsons JA, Shah BR, Mukerji G, Punthakee Z, Shulman R. An assessment of adaptation and fidelity in the implementation of an audit and feedback-based intervention to improve transition to adult type 1 diabetes care in Ontario, Canada. Implement Sci Commun. 2024 Mar 18;5(1):25. doi: 10.1186/s43058-024-00563-2. PMID 38500183
- [Derived] Shulman R, Zenlea I, Shah BR, Clarson C, Harrington J, Landry A, Punthakee Z, Palmert MR, Mukerji G, Austin PC, Parsons J, Ivers N. Testing an audit and feedback-based intervention to improve glycemic control after transfer to adult diabetes care: protocol for a quasi-experimental pre-post design with a control group. BMC Health Serv Res. 2019 Nov 25;19(1):885. doi: 10.1186/s12913-019-4690-0. PMID 31766999